CLINICAL TRIAL: NCT07071662
Title: Induction of Labor in Breech Presentation
Acronym: SIEGEC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0127
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Labor Induction at Term; Failure; Breech Presentation at Term
Keywords: labor induction; failure; breech presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaginal delivery
  Interventions: Other: delivery mode
- caesarean
  Interventions: Other: delivery mode

INTERVENTIONS:
Other: delivery mode — To observe the different modes of delivery and evaluate the characteristics of the patients as well as maternal and fetal well being in the post partum period.

SUMMARY:
Breech presenting fœtus were generally not offered a trial labor induction and were instead directed toward a cesarean section. This approach often led to obstetric complications for both the mother and the fetus.

This study aims to offer more labor inductions to patients with a fetus in breech presentation in order to avoid the mobidity and mortality associated with systematic cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* 34SA
* singleton
* consent for vaginal delivery
* breech presenting

Exclusion Criteria:

* -34SA
* minor
* twin pregnancy
* refusal of vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: patients with a fetus in breech presentation
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
number of vaginal delivery | day 1
Number of cesarean | day 1

SECONDARY OUTCOMES:
number of Endometrite | day 1
lactates value | day 1
Apgar value | day 1
Number of neonatology admission | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No